CLINICAL TRIAL: NCT05088005
Title: Prognostic Biomarkers of Mitochondrial and Oxidative Stress in Acute Carbon Monoxide Poisoning: Prospective Hyperbaric Oxygen Therapy Intervention Study
Brief Title: Prognostic Biomarkers in CO Poisoning
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: CO-new biomarkers
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Carbon Monoxide Poisoning; Hyperbaric Oxygenation; Biomarkers
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute CO poisoning: A diagnosis of CO poisoning was made according to medical history and carboxyhemoglobin >5% (>10% in smokers).
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Patients with any symptoms and signs were treated with HBO2. During the first HBO2, initial compression was performed to 2.8 atmospheres absolute (ATA) for 45 min, followed by 2.0 ATA for 60 min. If an additional HBO2 was possible within 24 h, then 2.0 ATA was administered for 90 min.

SUMMARY:
Mitochondrial and oxidative stress participate in the pathogenic mechanisms of carbon monoxide (CO)-induced toxicity. Thus, serum indicators of mitochondrial and oxidative stress could be useful for predicting neurocognitive prognosis of post-CO poisoning. This prospective observational study of consecutive patients requiring hyperbaric oxygen therapy (HBO2) for acute CO poisoning measured serum biomarkers of mitochondrial (growth differentiation factor 15 [GDF15]; fibroblast growth factor 21 [FGF21]) and oxidative (8-Oxo-2'-deoxyguanosine [8-OHdG] and malondialdehyde [MDA]) stresses at arrival at the emergency department (0 h), and at 24 h and 7 days after HBO2 completion. We evaluated neurocognitive outcomes using the Global Deterioration Scale (GDS; favorable [1-3 points] or poor [4-7 points] outcomes).

DETAILED DESCRIPTION:
Mitochondrial and oxidative stress participate in the pathogenic mechanisms of carbon monoxide (CO)-induced toxicity. Thus, serum indicators of mitochondrial and oxidative stress could be useful for predicting neurocognitive prognosis of post-CO poisoning.

This prospective observational study of consecutive patients requiring hyperbaric oxygen therapy (HBO2) for acute CO poisoning measured serum biomarkers of mitochondrial (growth differentiation factor 15 [GDF15]; fibroblast growth factor 21 [FGF21]) and oxidative (8-Oxo-2'-deoxyguanosine [8-OHdG] and malondialdehyde [MDA]) stresses at arrival at the emergency department (0 h), and at 24 h and 7 days after HBO2 completion. We evaluated neurocognitive outcomes using the Global Deterioration Scale (GDS; favorable [1-3 points] or poor [4-7 points] outcomes).

Levels of serum mitochondrial (GDF15 and FGF21) and oxidative stress (8-OHdG and MDA) biomarkers pre- and post-HBO2 were compared, to assess whether HBO2 reduced stress. In addition, we evaluated whether the blood test results correlated with the patient's neurocognitive prognosis at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* CO poisoned patients

Exclusion Criteria:

1. age < 19 years
2. a history of metabolic diseases
3. co-ingestion of drugs and alcohol, which may affect the biomarkers
4. discharge from the ED or transfer to another hospital
5. refusal to undergo HBO2
6. refusal to enroll in this study
7. lack of follow-up for assessing neurocognitive outcomes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CO poisoned patients
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Changes of serum biomarkers between pre-HBO2 and post HBO2 | At 1 day after HBO2
  Levels of serum mitochondrial (GDF15 and FGF21) and oxidative stress (8-OHdG and MDA) biomarkers pre- and post-HBO2 were compared, to assess whether HBO2 reduced stress.
Changes of serum biomarkers between pre-HBO2 and post HBO2 | At 7 days after HBO2
  Levels of serum mitochondrial (GDF15 and FGF21) and oxidative stress (8-OHdG and MDA) biomarkers pre- and post-HBO2 were compared, to assess whether HBO2 reduced stress.

SECONDARY OUTCOMES:
The prediction of poor neurocognitive outcome by serum biomarkers | At 1 month after CO exposure
  The prediction of serum biomarkers for the patient's neurocognitive prognosis at 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea